CLINICAL TRIAL: NCT02149641
Title: Phase II Study of Parotid Sparing IMRT for Nasopharyngeal Cancer
Brief Title: Parotid-sparing IMRT for Nasopharyngeal Cancer
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR2608
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Nasopharyngeal Cancers; Intensity Modulated Radiotherapy With Chemotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nasopharyngeal cancers: Intensitiy modulated radiotherapy with chemotherapy
  Interventions: Radiation: Intensity modulated radiotherapy with chemotherapy

INTERVENTIONS:
Radiation: Intensity modulated radiotherapy with chemotherapy

SUMMARY:
In the treatment of nasopharyngeal cancers, to determine the incidence of high grade (≥G2) subjective xerostomia at 1 year.

DETAILED DESCRIPTION:
The purpose of this study was to determine the feasibility in delivering induction chemotherapy and concomitant chemotherapy with IMRT in the treatment of locally advanced nasopharyngeal cancers and to determine the incidence of high grade (≥G2) subjective xerostomia at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* nasopharyngeal cancers

Exclusion Criteria:

* Patients <16 years old or with a previous malignancy other than non-melanomatous skin cancer were excluded

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: nasopharyngeal cancers
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2006-02; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
the incidence of ≥G2 xerostomia at 1 year using the subjective component LENTSOMA | 12 months

SECONDARY OUTCOMES:
Acute radiation toxicities | 0-3 months
Late radiation toxicities | 3-24 months
loco-regional disease-free survival (LRDFS), progression-free survival (PFS) and overall survival (OS) | 2 years
chemotherapy compliance and toxicities | 0-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Nutting, FRCR, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom